CLINICAL TRIAL: NCT00365495
Title: Influence of Physical Training on Mitochondrial Function in Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 022
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; physical training; mitochondrial function
MeSH Terms: conditions — Diabetes Mellitus, Type 2

INTERVENTIONS:
Procedure: Physical training (aerobic training)

SUMMARY:
Physical activity as treatment for patients with type 2 diabetes (T2D). Treatment of T2D is often done by medication, changing the diet and increased physical activity. It is well established that physical training has a positive effect on the pathology of T2D such as increased insulin sensitivity and reduced fasting plasma glucose (7) and blood lipids (15). It is also well known that in healthy subjects endurance training increases mitochondrial density, lipid oxidation during submaximal exercise, and results in a number of qualitative changes in the control of OXPHOS (24). However, the effect of physical training on the mitochondrial function in skeletal muscle of patients with T2D has not been investigated.

The purpose of this project is to investigate the effect of physical training on the mitochondrial respiratory function in muscles of patients with T2D. Skeletal muscle biopsies will be taken before and after 10 weeks of physical training in patients with T2D and matched control subjects. Mitochondria will be isolated from the muscle biopsies, and respiratory function, free radical production and UCP3 will be determined. Furthermore, measures of maximal oxygen consumption (VO2max), heart rate and capillary lactate concentrations and carbohydrate and lipid oxidation will be determined partly to verify an increased aerobic capacity and partly to investigate the changes in these factors in T2D patients.

ELIGIBILITY:
Inclusion Criteria:

* Male,
* BMI above 26,
* Age between 40 and 65,
* Living a sedentary lifestyle

Exclusion Criteria:

* Women
* BMI under 26
* Age under 40 and over 65
* Trained subjects Control subjects: relatives to type 2 diabetic patients, T2D trial subjects

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-08; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Mitochondrial respiratory measurements. The investigations are carried out by two rounds - one before Christmas and one after.

SECONDARY OUTCOMES:
VO2max
Lipid oxidation
muscle fiber type composition
muscle oxidative enzymes
mitochondrial-specific proteins (UCP3)
mitochondrial production of free oxygen radicals

CONTACTS AND LOCATIONS:
Overall Officials: Martin Mogensen, PhD student, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark and Odense University Hospital, Odense, Denmark